CLINICAL TRIAL: NCT04349371
Title: Chloroquine (CQ) Prophylaxis for Health Care Workers at Risk for COVID
Brief Title: Saved From COVID-19 - Chloroquine (CQ) Prophylaxis for Health Care Workers at Risk for COVID
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment.
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Anca Askanase, Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAS9992
Record Dates: First submitted 2020-04-12; First posted 2020-04-16 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: COVID; Coronavirus Infection
Keywords: SARS-CoV-2; Coronavirus
MeSH Terms: conditions — Coronavirus Infections | interventions — Chloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CQ group (Experimental): Participants will receive CQ supply for 3 months. Patients will receive a supply of 36 -- 250 mg tabs or placebo that will last 3 months (enough for taking two tabs of 250mg for every day for one week and then two tabs of 250mg for 1 day a week thereafter for study duration of 3 months). Subjects with severe GI intolerance can take 1 tablet of 250mg daily for the first week and 1 tablet per week for the remainder of the 3 month study duration. Patients will attend 1 in person visits (month 0) and an additional visit during month 3 if possible with the physician where they will be evaluated for safety assessments including vital signs, physical exams, blood collection, and assessment of endpoints. During month 1, 2, and 3 participants will be followed up regarding concomitant medications and adverse events over the phone call.
  Interventions: Drug: Chloroquine
- Placebo group (Placebo Comparator): Participants will receive placebo supply for 3 months. Patients will attend 1 in person visits (month 0) and an additional visit during month 3 if possible with the physician where they will be evaluated for safety assessments including vital signs, physical exams, blood collection, and assessment of endpoints. During month 1, 2, and 3 participants will be followed up regarding concomitant medications and adverse events over the phone call.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Chloroquine — Subjects will take two tabs of 250mg for every day for one week and then two tabs of 250mg for 1 day a week thereafter for study duration of 3 months). Subjects with severe GI intolerance can take 1 tablet of 250mg daily for the first week and 1 tablet per week for the remainder of the 3 month study duration.
  Other Names: CQ
  Arms: CQ group
Drug: Placebo oral tablet — Subjects will take two tabs of placebo for every day for one week and then two tabs of placebo for 1 day a week thereafter for study duration of 3 months).
  Other Names: Placebo pill
  Arms: Placebo group

SUMMARY:
The primary objective is to determine the clinical efficacy of Chloroquine (CQ) in health care workers with moderate to high risk of exposure to COVID-19 in preventing symptomatic COVID-19 infections. Secondary endpoints will explore the efficacy of CQ in preventing any infection as defined by seroconversion to positive anti-COVID antibody status.

DETAILED DESCRIPTION:
Chloroquine (CQ) phosphate is an immunomodulatory drug that has been approved by the FDA for prophylaxis of and treatment of malaria, treatment of lupus erythematosus, and treatment of rheumatoid arthritis. Anecdotal data and in-vitro studies suggests potential benefit of chloroquine in treating COVID-19 patients. The use of CQ to treat COVID-19 patients have been demonstrated to be effective in inhibiting severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The use of CQ in health care workers with moderate to high risk of exposure to COVID-19 in could prevent symptomatic COVID 19 infections. 350 participants will be randomized (like a flip of a coin) to a 3 month chloroquine versus an identical course of placebo. A placebo is a sugar pill which has no active ingredient. will attend one in person visit during month 0 for screening and randomization, and if possible during the last visit at month 3. During month 1 and 2 the in person visits are optional and the PI can follow up with subjects through telemedicine or phone call. Informed consent, inclusion/exclusion criteria, demographic, medical/ disease history/ comorbidity/ medical records review, prior/ concomitant meds and procedures, and adverse events will be collected from patient during screening visit 1 (month 0). Limited physical assessment, vitals, blood serum, investigational product compliance review, assessment of adverse events, serious adverse events, adverse events of special interest, and endpoint assessments are also collected during visit 1. Prior/concomitant medications and procedures, adverse events, study drug compliance review, adverse events of special interest, adverse events of special interest and endpoint assessments will be reviewed at every visit. Blood serum will be collected during visits 1 (month 0) and at visit 4 (month 3) if subject can come to the visit physically. By the end of the study, the investigators hope that there is decrease of symptomatic illness in at risk healthcare workers and a decrease in symptomatic COVID infection.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years,
2. Employment by New York Presbyterian Hospital
3. Clear assignment to areas of the hospital that involve patient contact and possible exposures for at least 2 days a week >/= 8 hours a day

Exclusion Criteria:

1. Individuals who are taking CQ for other indications
2. New use of NSAIDs
3. High risk background medications not limited to immunosuppressive regimens, steroids, anti-B cell therapies, anti-cytokine therapies, chemotherapies, Janus Kinase (JAK)-inhibitors
4. Individuals with a history of retinopathy that would contraindicate the use of CQ
5. Known allergy to CQ or chloroquine
6. Known QT prolongation and torsades de point
7. Individuals who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anca Askanase, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center/NYP, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated before participants could be assigned to any Arm. There were 5 participants who signed informed consent form: 3 participants withdrew, and 2 participants did not proceed due to study termination.
Groups:
- CQ Group: The study was terminated before participants could be assigned to any Arm. Per protocol, participants will receive CQ supply for 3 months.
- Placebo Group: The study was terminated before participants could be assigned to any Arm. Per protocol, participants will receive placebo supply for 3 months.
Period: Overall Study
Arm/Group | CQ Group | Placebo Group
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated before participants could be assigned to any Arm.
Groups:
- CQ and Placebo Group: Participants will receive CQ or placebo supply for 3 months.
Arm/Group | CQ and Placebo Group
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Number of Healthcare Workers With Symptomatic COVID Infections
Description: Diagnosis is based on symptoms of COVID-19 and confirmatory anti-COVID antibodies and when available, COVID-19 PCR. This is to determine/measure the clinical efficacy of CQ in healthcare workers.
Time Frame: Up to 3 months
Population: The study was terminated before participants could be assigned to any Arm. Data was therefore not collected or analyzed.
Groups:
- CQ and Placebo Group: Participants will receive CQ or placebo supply for 3 months.
  The study was terminated before participants could be assigned to any Arm.
Arm/Group | CQ and Placebo Group
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Workers and Patients With Infections
Description: This is to measure the efficacy of CQ in preventing any infection as defined by seroconversion to positive anti-COVID antibody status.
  The number of severe illnesses in at risk healthcare workers and patients with adverse events grade 3 or higher and GI intolerance will be tallied.
Time Frame: 3 months
Population: The study was terminated before participants could be assigned to any Arm. Data was therefore not collected or analyzed.
Arm/Group | CQ and Placebo Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 3 months
Description: The study was terminated before participants could be assigned to any Arm, therefore Adverse Events cannot be reported per Arm.
Arm/Group | CQ and Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
Study was stopped early due to poor enrollment. Data was not collected and therefore not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT04349371/Prot_SAP_000.pdf